CLINICAL TRIAL: NCT05826561
Title: Developing a Childhood Asthma Risk Passive Digital Marker
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: NIH funding was terminated due to new agency priorities.
Sponsor: Indiana University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Arthur H. Owora, MPH, PhD, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 15873; K01HL166436 (NIH)
Record Dates: First submitted 2023-04-12; First posted 2023-04-24 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Asthma
Keywords: Pediatric Asthma; Early Detection; Screening; Passive Digital Marker; Risk Factors

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Clinicians - post test only (No Intervention): N=25 control pediatric clinicians, who will receive the post test only. Each clinician will be presented with 10 randomly selected vignettes of 10 children [5 with and 5 without asthma] and asked to provide a prediction of a child's asthma risk at 6-10 years.
- PDM Intervention Clinicians - post test only (Experimental): N=25 intervention pediatric clinicians, who will receive the post test only. Using the PDM, each clinician will be presented with 10 randomly selected vignettes of 10 children [5 with and 5 without asthma] and asked to provide a prediction of a child's asthma risk at 6-10 years.
  Interventions: Other: Childhood Asthma Passive Digital Marker
- Control Clinicians - pre and post test (No Intervention): N=25 control pediatric clinicians, who will receive the pre and post test. Each clinician will be presented with 10 randomly selected vignettes of 10 children [5 with and 5 without asthma] and asked to provide a prediction of a child's asthma risk at 6-10 years.
- PDM Intervention Clinicians - pre and post test (Active Comparator): N=25 intervention pediatric clinicians, who will receive the pre and post test. Using the PDM, each clinician will be presented with 10 randomly selected vignettes of 10 children [5 with and 5 without asthma] and asked to provide a prediction of a child's asthma risk at 6-10 years.
  Interventions: Other: Childhood Asthma Passive Digital Marker

INTERVENTIONS:
Other: Childhood Asthma Passive Digital Marker — A childhood asthma Passive Digital Marker (PDM) is an ML algorithm that is able to retrieve and synthesize pre-existing "passively" collected mother/child dyad prognostic data in "digital" electronic health record (EHR) to provide an objective and quantifiable "marker" of a child's risk (probability) and associated pathophysiological phenotype to inform clinician decision-making at point-of-care.
  Other Names: Passive Screening Test (PDM)
  Arms: PDM Intervention Clinicians - post test only; PDM Intervention Clinicians - pre and post test

SUMMARY:
Underdiagnosis and undertreatment is a major problem in childhood asthma management, especially in preschool-aged children. Current prognostic approaches using risk-score based tools have poor-to-modest accuracy, are impractical, and have limited evidence of efficacy in clinical settings and hence are not widely used in practice.

The objective of the study is to determine the usability, acceptability, feasibility, and preliminary efficacy of the childhood asthma passive digital marker (PDM) among pediatricians. The study will include practicing pediatricians within the IU Health Network.

ELIGIBILITY:
Inclusion Criteria:

• Practicing pediatricians within the IU Health Network

Exclusion Criteria:

• Non-practicing pediatricians within the IU Health Network

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Perceived PDM acceptance | 8 to 12 months
  Perceived PDM acceptance will be measured using a Behavioral Intention scale (BIS).
Perceived PDM usability | 8 to 12 months
  Perceived Usability will be measured using a modified Simplified System Usability Scale (SUS).
Study feasibility | 8 to 12 months
  Percent of successful study enrollment of eligible clinicians (>80%)

SECONDARY OUTCOMES:
Prognostic accuracy | 3 to 12 months
  % correct clinician predictions at pre and post test

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Indianapolis, Indiana, United States